CLINICAL TRIAL: NCT06615934
Title: Comparing the Effects of Aerobic and Resistance Exercises With Routine Physiotherapy in Inpatients Immediately After Liver Transplantation on Muscle Strength, Functional and Aerobic Capacity, and Blood Biomarkers
Brief Title: Effects of Aerobic and Resistance Exercises on Inpatients Liver Transplantation Recipients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mohammad Javaherian, Dr. Mohammad Javaherian, Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 65214
Record Dates: First submitted 2024-05-06; First posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Liver Transplant Disorder; Liver Transplant; Complications; End-stage Liver Disease
Keywords: physiotherapy; aerobic exercise; resistance exercise; liver transplant recipients
MeSH Terms: conditions — End Stage Liver Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic and resistance exercise (Experimental): respiratory physiotherapy + aerobic and resistance exercise therapy
  Interventions: Other: Aerobic and resistance exercise
- Respiratory physiotherapy (Active Comparator): respiratory physiotherapy alone
  Interventions: Other: Aerobic and resistance exercise; Other: Respiratory physiotherapy

INTERVENTIONS:
Other: Aerobic and resistance exercise — From the first day of transplantation in the ICU until 10 days after transfer to the ward or discharge from the hospital, if needed, the patients of the group will undergo respiratory physiotherapy once a day. The process of this program includes patient assessment, clinical decision-making, and implementation of therapeutic interventions.
  The interventions of the therapeutic exercise group are divided into three phases:
  1. From the time the patient enters the ICU until the time of extubation;
  2. From the time of extubation to the time of transfer to the ward;
  3. Duration of the patient's stay in the ward.
Other: Respiratory physiotherapy — The participants of this group will receive respiratory physiotherapy daily after transplant until discharge.
  Arms: Respiratory physiotherapy

SUMMARY:
The prevalence of chronic liver disease and primary liver cancer is still increasing on a global scale, and so are their associated deaths.

Compared to other diseases, death from liver disease often means premature death, because two-thirds of the lives lost are working years.

Liver transplantation (LT) is an important and life-saving treatment option for the treatment of congenital metabolic disorders, acute liver failure, end-stage chronic liver disease (ESLD) and primary liver cancers.

Modern liver transplantation is characterized by significant improvements in post-transplant patient survival, graft survival, and quality of life.

Impaired physical fitness of patients with end-stage liver disease often persists after liver transplantation and compromises post-transplant recovery.

Prior to liver transplantation, excess ammonia taken up by skeletal muscle is a major metabolic driver of muscle wasting in end-stage liver disease and mainly inhibits the mTOR signaling pathway that supports muscle protein synthesis.

Because excess ammonia is no longer present after transplantation, recovery of muscle mass and function can be expected in patients. However, immunosuppression with calcineurin inhibitors that inhibit the mTOR signaling pathway may improve lethal length.

It is also thought that post-transplant treatment regimens contribute to delayed recovery of decreased bone mineral density and increased fracture risk.

Greater muscle mass, as measured by creatinine clearance at 1 year after transplantation, was associated with longer recipient and allograft survival.

The results of previous studies indicate low cardiovascular fitness in patients after liver transplantation.

Since after liver transplantation, cardiovascular diseases cause 19 to 42% of deaths not related to the liver, performing aerobic exercises to obtain and maintain cardiovascular fitness after liver transplantation can reduce the mortality rate. After transplanting, reduced significantly.

Considering the important role of the immune system in transplant rejection, the safety of sports training is very important in terms of not over-activating the immune system and endangering the life of the transplanted tissue. In previous studies related to exercise and immune system activity and inflammatory cytokines after transplantation, it has been shown that moderate exercise including aerobic and resistance exercises can inhibit inflammatory cytokines and have beneficial effects on the immune system.

High levels of tumor necrosis factor-alpha (TNF-α) in the period after transplant surgery are associated with an increased risk of transplant rejection.

Aerobic exercise reduces levels of inflammatory cytokine TNF-α and markers of liver function in patients with chronic liver diseases.

According to this evidence, it seems that doing sports exercises is effective in reducing the risk of transplant rejection and modulating the patient's immune system. Acute graft rejection occurs days to weeks after transplantation. The immune system can see the transplanted organ as foreign and attack it, destroy it and lead to transplant rejection.

Considering the mentioned benefits of exercise therapy after liver transplantation, it is possible that the early start of exercise therapy in the hospitalization phase leads to a reduction in the risk of transplant rejection and improvement of allograft residues in patients after liver transplantation.

Considering that the current evidence shows that there is no use of a specific rehabilitation protocol in the hospitalization phase of patients after liver transplantation, we intend to evaluate its effects with changes in the common physiotherapy program in these departments according to the specific conditions of these patients. In other words, despite the acceptable therapeutic effects, the use of a combined protocol of aerobic and resistance exercises in the hospitalization phase of these patients has not been reported so far.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who undergo elective surgery after the approval of the liver transplant commission.
2. Having an underlying liver disease with metabolic disorder (as determined by the Liver Transplantation Commission)
3. Absence of transplantation of other organs
4. No re-transplantation of the liver
5. Age more than 18 years
6. Ability to participate in initial evaluations
7. Patient's ability to understand questionnaire questions

Exclusion Criteria:

1. The patient's lack of satisfaction with continuing cooperation for any reason
2. Re-transplantation up to 3 months after discharge
3. Facing the patient with early allograft dysfunction or primary nonfunction
4. Encountering the criteria of non-implementation of the intervention during 50% of the days of stay in the hospital or more
5. Patients with Postoperative respiratory failure (Extubation > 48 hours)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2024-12-15 (Estimated); Study Completion 2025-01-15 (Estimated)

PRIMARY OUTCOMES:
Six-minute walk test | Before transplantation (Day 0), after 10 sessions (An average three weeks), and three months after discharge (An average, 16 weeks)
  The distance traveled by each patient after 6 minutes of walking will be calculated using a laser meter.

SECONDARY OUTCOMES:
Muscle Strength | Before transplantation (Day 0), after 10 sessions (An average three weeks), and three months after discharge (An average, 16 weeks)
  Shoulder abductor, elbow flexor, hip flexor, and knee extensor muscle groups of the dominant side
Health-related quality of life | Before transplantation (Day 0), after 10 sessions (An average three weeks), and three months after discharge (An average, 16 weeks)
  Using the short form of the 36-question health-related quality of life questionnaire (SF-36) The scores of SF-36 questionnaire are presented from 0 to 100 which higher scores indicates better quality of life.
Health-related quality of life (PLTQ) | Before transplantation (Day 0), after 10 sessions (An average three weeks), and three months after discharge (An average, 16 weeks)
  Using the post-Liver Transplant Quality of Life questionnaire (PLTQ). The PLTQ scores are presented from 0 to 32 which higher score indicated better level of quality of life.
Cardiopulmonary exercise test | Before transplantation (Day 0), after 10 sessions (An average three weeks), and three months after discharge (An average, 16 weeks)
  The process of performing this test will be based on the CPET guidelines of the American Heart Association and according to the modified Bruce protocol. The results of this test will be maximum oxygen consumption (Vo2 max) and anaerobic threshold (AT), which is in mL/kg/min.
The level of Urea | Before transplantation (Day 0), after 10 sessions (An average three weeks), and three months after discharge (An average, 16 weeks)
  The serum level of urea which will be analyzed from blood samples and can indicate the function of liver and kidney.
The level of Creatinine | Before transplantation (Day 0), after 10 sessions (An average three weeks), and three months after discharge (An average, 16 weeks)
  The serum level of creatinine which will be analyzed from blood samples and can indicate the function of liver and kidney.
The level of Interleukin-6 | Before transplantation (Day 0), after 10 sessions (An average three weeks), and three months after discharge (An average, 16 weeks)
  The serum level of interleukin-6 which indicated the level of inflammation of internal organs.
The level of Tumor Necrosis Factor-alpha | Before transplantation (Day 0), after 10 sessions (An average three weeks), and three months after discharge (An average, 16 weeks)
  The serum level of Tumor Necrosis Factor-alpha (TNF-alpha) which indicates diverse range of signaling events within cells and level of cell necrosis.

CONTACTS AND LOCATIONS:
Overall Officials: Behrouz Attarbashi Moghadam, Ph.D., Principal Investigator — Department of Physiotherapy,Tehran University of Medical Sciences,Tehran,Iran.
Locations (1):
- Liver Transplantation Research Center, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Yes
Researchers can access the study protocol and limited data from some participants (anonymous) after sending their requests and approved proposal with ethical committee confirmation.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Six months after publishing the final article of the study.